CLINICAL TRIAL: NCT05493163
Title: A Multicentre, Randomized Trial of Catheter-directed Thrombolysis in Intermediate-high Risk Acute Pulmonary Embolism (PRAGUE-26)
Brief Title: Catheter-directed Thrombolysis in Intermediate-high Risk Acute Pulmonary Embolism
Acronym: PRAGUE-26
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Collaborators: Charles University, Czech Republic (Other); University Hospital Ostrava (Other); University Hospital Olomouc (Other); University Hospital Brno (Unknown); St. Anne´s University Hospital Brno (Unknown); General University Hospital, Prague (Other); University Hospital Pilsen (Other); Pardubice Hospital (Unknown)
Responsible Party: Principal Investigator, Viktor Kocka, Chief Interventional cardiologist, Faculty Hospital Kralovske Vinohrady
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRAGUE-26; 2022-002218-18 (EudraCT Number)
Record Dates: First submitted 2022-07-30; First posted 2022-08-09 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Embolism
Keywords: Acute Pulmonary Embolism; Local Thrombolysis; Catheter-Directed Thrombolysis; Intermediate-High Risk
MeSH Terms: conditions — Pulmonary Embolism | interventions — Fibrinolytic Agents

STUDY DESIGN:
Intervention Model Description: Prospective, multicentre, randomized, active-controlled, unblinded, parallel-group study to evaluate clinical outcomes in patients with intermediate-high risk acute PE undergoing CDT in comparison to standard anticoagulation therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catheter-Directed Thrombolysis (Experimental): Venous access should be obtained under ultrasound guidance (via the common femoral vein). The use of a double-lumen 8-Fr introducer (single access site) or two 4-Fr introducers (two ipsilateral access sites) is at the discretion of the operator.
  After each thrombolytic catheter placement into left and/or right pulmonary artery, a subsequent bolus of 1mg of Alteplase (Actilyse, Boehringer Ingelheim)/catheter is administered, followed by continuous infusion at 1 mg/h/catheter for 9 h (total dose 10mg for unilateral and 20mg for bilateral PE).
  Intravenous unfractionated heparin is continued to a target activated partial thromboplastin time (aPTT) of 50-60 s. After the end of local thrombolysis, the catheters are removed and anticoagulation with unfractionated heparin continues.
  Interventions: Drug: Thrombolytic
- Standard Anticoagulation (Active Comparator): Before randomization, all patients are treated with intravenous unfractionated heparin (to a target aPTT of 70-90 s) or subcutaneous LMWH (the full therapeutic dose). For patients in the CDT group, the anticoagulation treatment was is described above; among CDT patients who received LMWH, the procedure should be postponed for 8 h after the last dose of LMWH. Patients in the standard care group continue therapeutic anticoagulation with either unfractionated heparin or LMWH. Subsequent change for oral anticoagulation is at the discretion of the treating physician (not earlier than 24 hours post-randomization).
  Interventions: Drug: Standard anticoagulation

INTERVENTIONS:
Drug: Thrombolytic — Local, catheter-directed thrombolysis with a total dose of 10mg per affected lung administered over 9 hours.
  Arms: Catheter-Directed Thrombolysis
Drug: Standard anticoagulation — Standard anticoagulation therapy of acute pulmonary embolism.
  Arms: Standard Anticoagulation

SUMMARY:
Background: Intermediate-high risk acute pulmonary embolism (PE) remains associated with substantial mortality despite standard anticoagulation therapy. Previous efforts to decrease mortality in these patients via administration of systemic thrombolysis have failed due to an increased rate of major bleeding complications. Catheter-directed thrombolysis (CDT) has already shown some promising results in terms of efficacy and safety, including the results of our randomized pilot study. However, large randomized trials with clinical endpoints comparing catheter-directed local thrombolysis versus standard anticoagulation therapy are still lacking, thus the treatment of intermediate-high risk acute PE patients has not changed for decades. Hypothesis: Catheter-directed local thrombolysis is superior to standard anticoagulation therapy in the treatment of intermediate-high risk acute pulmonary embolism, with no additional safety concerns. Statistical considerations: Estimated incidence of the primary endpoint of 1.5% in the CDT group and 6.0% in the standard anticoagulation group, 80% power for each arm with a 2-sided alpha of 0.05. Five hundred fifty-eight should provide the requisite number of events. Statistical Analysis - Intention to Treat. Methods and Results: A Multicentre, Randomized Trial of Catheter-directed thrombolysis in intermediate-high risk acute pulmonary embolism (PRAGUE-26) is a noncommercial, multicentre, randomized, controlled parallel-group comparison trial. The trial plans to include 558 patients with intermediate-high risk acute PE. Patients will be randomized in a 1:1 ratio to CDT or to standard anticoagulation therapy. The primary outcome of the study is a clinical composite of all-cause mortality, PE recurrence or cardiorespiratory decompensation, within 7 days of randomization. Secondary objectives cover all bleeding complications, functional and patient-reported outcomes over a follow-up period of 24 months and cost-effectiveness analysis.

DETAILED DESCRIPTION:
1. Introduction Intermediate-high risk acute pulmonary embolism (PE) remains associated with substantial mortality despite standard anticoagulation therapy [1]. Previous efforts to decrease mortality in these patients via administration of systemic thrombolysis have failed; such treatments were associated with major bleeding complications [2,3]. Catheter-directed thrombolysis (CDT) has already shown some promising results; effectively reducing right ventricle (RV) overload, decreasing systolic pulmonary artery pressure (sPAP), and reducing pulmonary thrombotic burden while remaining safe for the patient (i.e., not increasing the rate of intra-cranial or life-threatening bleeding complications) [4-7]. There are currently two main treatment options - ultrasound-assisted local thrombolysis (USAT) or simple catheter-directed local thrombolysis (i.e., without ultrasound facilitation). The USAT has yielded promising results, but is expensive and thus infrequently used. Simple CDT has shown similar efficacy compared to USAT [8] and represents a low-cost alternative. Unfortunately, randomized trials with clinical endpoints are still lacking [9].

   Investigators have performed a first randomized pilot trial of catheter-directed thrombolysis or standard anticoagulation therapy in patients with intermediate-high acute pulmonary embolism [10]. In this randomized trial, a safe and simple method of CDT was introduced. Efficacy in terms of RV function improvement (RV/LV ratio reduction) and systolic pulmonary artery pressure reduction compared to standard anticoagulation therapy was demonstrated, with no safety concerns.

   Recently, enrolment in HI-PEITHO Trial (sponsored by Boston Scientific Corporation) has begun investigating the clinical outcomes of intermediate-high risk acute PE patients undergoing USAT (EKOS system) plus anticoagulation therapy compared to anticoagulation therapy alone (NCT04790370) [11].

   However, there is currently no randomized trial investigating the clinical outcomes in patients undergoing simple CDT plus anticoagulation compared to anticoagulation therapy alone.
2. Study objectives The purpose of this study is to investigate clinical outcomes in patients with intermediate-high risk acute PE undergoing catheter-directed (local) thrombolysis compared to standard anticoagulation therapy.
3. Study design Prospective, multicentre, randomized, active-controlled, unblinded, parallel-group study to evaluate clinical outcomes in patients with intermediate-high risk acute PE undergoing CDT in comparison to standard anticoagulation therapy.

   3.1 Randomization A web-based randomization software will be used for the randomization with a ratio of 1:1. Randomization into treatment groups will be stratified by the following criteria: age, gender, uni- or bilateral acute PE*, time from the diagnosis of acute PE (diagnostic CT angiography), direct admission to tertiary care cardio centre.

   * bilateral acute PE definition - a perfusion defect in at least one main or one lobar pulmonary artery simultaneously in the left and in the right lung evident on CT angiography.

   3.2 Screening, randomization and treatment All patients will undergo routine clinical evaluation and standard of care testing (CT angiography, transthoracic echocardiography, laboratory testing) for the diagnosis and risk stratification of acute PE.

   There is no time limit from the CT angiography confirmed diagnosis of intermediate-high risk acute PE to randomization, but investigators should take measures to minimize the duration of time to randomization into the study.

   Patients meeting all inclusion criteria and not meeting any of exclusion criteria will be randomized on Day 1, which will be the day of CDT procedure in patients allocated into the CDT group. The other patients will continue standard anticoagulation therapy as a standard of care.

   Patients will be assessed for AEs, SAEs for 12 months post-randomization. Patients will be invited for out-patient visit at the time of 30 days (± 3 days), 12 months (± 14 days) and 24 months (± 14 days) post-randomization.

   When the prespecified number of adjudicated clinical endpoint events have been reached, all centres will be notified by Principal investigator´s study team.

   3.3. Data Safety Monitoring Board Data safety monitoring board (DSMB) will monitor the progress of the study and ensure that the safety of patients in the study is not compromised. The DSMB will review accumulating data on regular basis. There will be an interim analysis at 50% and 75% of enrolled number of patients. Based on review of clinical events and safety events the DSMB will make recommendations on the continuation of the study or may recommend early termination of the study.
4. Study endpoints see next section
5. Statistics Based on the PEITHO study (primary composite endpoint of death or hemodynamic collapse with incidence of 5.6% in standard arm) [3], based on the study published by Becattini (early mortality of 6.0-7.7%) [1] and based on randomized pilot study [10] the incidence of primary composite endpoint of 1.5% in the CDT group and 6.0% in the standard care group was estimated. Power calculation is shown below.

   1. Incidence, Group CDT 1.5% N=279
   2. Incidence, Group Standard anticoagulation 6% N=279 With Alpha=0.05, Beta=0.2 a total predicted number of patients is 558. Power calculation - Sample Size Calculator. https://clincalc.com/stats/samplesize.aspx
6. Inclusion and Exclusion criteria see next section
7. Procedures and Assessments Eligible patients may only be included in the study after providing written (witnessed, where required by law or regulation) Institutional Ethics Committee approved informed consent.

   7.1 Catheter-directed thrombolysis and anticoagulation All interventional procedures should be performed as soon as possible post-randomization (max. within 3 hours). After previous exclusion of deep vein thrombosis via ultrasound or CTA, venous access should be obtained under ultrasound guidance (via the common femoral vein). The use of double-lumen 8-Fr introducer (single access site) or two 4-Fr introducers (two ipsilateral access sites) is at the discretion of the operator. Subsequent steps of the procedure (procedure methodology) were described in previously published pilot study [10].

   After each catheter placement, subsequent bolus of 1mg of Alteplase (Actilyse, Boehringer Ingelheim)/catheter is administered, followed by continuous infusion at 1 mg/h/catheter for 9 h (total dose 10mg for unilateral and 20mg for bilateral PE). This dosing of Alteplase is significantly lower than the standard guideline-based dose of 100mg which is recommended for patients with high-risk PE with shock or hypotension. All studies with local thrombolysis have used similarly low dose and it is reassuring that the risk of intracranial or life-threatening bleeding does not seem increased. [4-7] One small study studied the dosing and duration of Alteplase infusion, the total dose ranged from 8 to 24mg and a higher dose seemed numerically more effective.[7] These data form the scientific basis for the selection of Alteplase dose. Independently, the recently initiated multicentre HI-PEITHO study of ultrasound-assisted local thrombolysis has opted for very similar dosing of 9mg for unilateral and 18mg for bilateral PE.[11] Intravenous unfractionated heparin is continued to a target activated partial thromboplastin time (aPTT) of 50-60 s. After the end of local thrombolysis, the catheters are removed and anticoagulation with unfractionated heparin (without a bolus) is continued to a target aPTT of 70-90 s. The 8-Fr introducer (or two 4-Fr introducers) is removed from the femoral vein 60 min after the end of Alteplase infusion, and the access site is manually compressed for 10 min.

   Anticoagulation. Before randomization, all patients are treated by intravenous unfractionated heparin (to a target aPTT of 70-90 s) or subcutaneous LMWH (the full therapeutic dose). For patients in the CDT group, the anticoagulation treatment was is described above; among CDT patients who received LMWH, the procedure should be postponed for 8 h after the last dose of LMWH. Patients in the standard care group continue therapeutic anticoagulation with either unfractionated heparin or LMWH. Subsequent change for oral anticoagulation is at the discretion of treating physician (not earlier than 24 hours post-randomization).

   7.2 Other procedures CT angiography (CTA). Diagnostic CTA is a component of routine clinical care. No other CTA is required unless clinically indicated (e.g., acute PE recurrence, etc.).

   Transthoracic echocardiography (TTE). Transthoracic echocardiography is a component of routine clinical care. The second TTE will be performed on Day 1 (max. within 3 hours post-randomization) and the third TTE will be performed 24 (± 3 hours) post-randomization. There will be another echocardiographic assessment during out-patient visits (at 30 days, 12 months and 24 months). Standard measurements will be performed in accordance with the European Society of Cardiology recommendations [12,13]. The subannular RV/LV ratio will be derived as suggested by the ULTIMA study [6].

   Laboratory tests. Standard laboratory tests (biochemistry, hematology, coagulation) are a component of routine clinical care. In patients undergoing the CDT procedure, additional laboratory tests (blood count, aPTT, INR, fibrinogen) are recommended 6 hours after Alteplase infusion initiation.

   Functional assessment. Patients' functional status will be assessed at prespecified time frames using a WHO functional class classification, 6-Minute Walk Test, and EQ-5D scale.

   7.3 Concomitant medication, prohibited medication Patients strictly follow the protocol on anticoagulation therapy as described above. All other anticoagulants (e.g., warfarin, fondaparinux, edoxaban, etc.) than unfractionated heparin or low-molecular-weight heparin are prohibited during first 24 hours post-randomization. The only exception is a rescue thrombolysis in case of cardiorespiratory decompensation. Patients with the prior use of antiplatelet drugs may continue with antiplatelet treatment if clinically indicated. In case of bleeding event the treatment can be modified and other necessary medication can be administered to solve adverse events.
8. Study Assessment Schedule will be provided in the Protocol file
9. Regulatory issues This study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki, as well as national legal and regulatory requirements.

Study-related correspondence, subject records, consent forms, and source documents are to be maintained on file by the trial site. Records of each subject's participation in the trial must be maintained for no less than a period of two (2) years after trial closure and submission of the final report to the EC, or longer as dictated by local regulations/local regulatory authority.

Changes in the protocol affecting the study outcome are made only by written amendment agreed upon by the trial Sponsor, the Ethical Committee (EC), and if pertinent, any other applicable regulatory agency/authority. As appropriate, the trial Sponsor will submit changes in the protocol and investigators will obtain EC re-approval. A report of withdrawal of EC approval must be submitted to the trial Sponsor within five (5) business days. Any major revisions to the protocol, must be approved by trial Sponsor, by the EC and local regulatory authority.

A final clinical report shall be compiled once data collection is complete. Such reports include all information required and outlined in this protocol. The final report will be provided to ECs and other regulatory agencies as per applicable laws. The final clinical report will be filed in the clinical trial databases.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years and not over 80 years.
2. Computed tomography angiography (CTA)-verified proximal* PE AND symptom onset < 14 days prior.
3. Intermediate-high risk PE with a SPESI score ≥ 1 AND RV dysfunction** AND an elevated biomarker *** (hs-troponin or NT-proBNP) level.
4. Signed informed consent.

Exclusion Criteria:

1. Active clinically significant bleeding.
2. Any haemorrhagic stroke OR a recent (< 6 months) ischaemic stroke/transient ischaemic attack.
3. Recent (< 3 months) cranial trauma OR another active intracranial/intraspinal process.
4. Major surgery within 7 days prior.
5. Active malignancy OR other severe illness with expected survival < 2 years.
6. Haemoglobin level < 80 g/L; international normalised ratio > 2.0, platelet count ≤ 100 x 109; creatinine level > 200 µmol/L.
7. Pregnant or breastfeeding, fertility without previous exclusion of gravidity.
8. Allergic to thrombolytics or heparin or low-molecular-weight heparin (LMWH), contrast allergy, a history of heparin-induced thrombocytopenia.
9. Floating thrombi in transit through a patent foramen ovale.
10. Participation in another clinical trial.

    * A perfusion defect in at least one main or one lobar pulmonary artery is evident on CTA.

      * RV/LV ratio ≥ 0.9 on transthoracic echocardiography or CTA. *** hs-troponin I (TnI) > 53 ng/L (men) or > 34 ng/L (women); NT-proBNP level > 600 pg/mL.

SPESI - Simplified Pulmonary Embolism Severity Index.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | 7 days
  Combined; clinical composite of any of the following parameters within 7 days of randomization
  1. All-cause mortality
  2. PE recurrence (non-fatal symptomatic and objectively confirmed recurrence of PE by repeated CTA)
  3. Cardiorespiratory decompensation or collapse* * Defined as at least one of following criteria:
     1. cardiac arrest or need for CPR at any time between randomization and day 7;
     2. signs of shock;
     3. placement on extracorporeal membrane oxygenation (ECMO);
     4. intubation, or initiation of non-invasive mechanical ventilation at any time between randomization and day 7;
     5. National Early Warning Score (NEWS) of 9 or higher, between 24 hours and 7 days after randomization, confirmed on consecutive measurements taken twice, 15 minutes apart.

SECONDARY OUTCOMES:
Secondary endpoints | 7 days to 24 months
  All-cause mortality
Secondary endpoints | 7 days to 24 months
  PE recurrence (non-fatal symptomatic and objectively confirmed recurrence of PE by repeated CTA)
Secondary endpoints | 7 days
  Cardiorespiratory decompensation or collapse*
  * Defined as at least one of following criteria:
  1. cardiac arrest or need for CPR at any time between randomization and day 7;
  2. signs of shock;
  3. placement on extracorporeal membrane oxygenation (ECMO);
  4. intubation, or initiation of non-invasive mechanical ventilation at any time between randomization and day 7;
  5. National Early Warning Score (NEWS) of 9 or higher, between 24 hours and 7 days after randomization, confirmed on consecutive measurements taken twice, 15 minutes apart.
Secondary endpoints | 30 days
  First-line therapy failure**
  ** Defined as administration of systemic thrombolysis during first (index) hospitalization for acute PE.
Secondary endpoints | 7 and 30 days
  Ischemic or haemorrhagic stroke
Secondary endpoints | 12 months
  Serious adverse events
Secondary endpoints | 30 days
  Duration of hospitalization for the index acute PE event (Time from admission to discharge from hospital)
Secondary endpoints | 30 days
  Duration of stay at the intensive, intermediate or coronary care unit during hospitalization for the index acute PE event (Time from admission to discharge from ICU, intermediate, or CCU)
Secondary endpoints | 30 days
  Hospitalization cost (cost-effectiveness analysis)
Secondary endpoints | 30 days
  GUSTO major (moderate and severe) bleeding
Secondary endpoints | 30 days
  International Society on Thrombosis and Hemostasis (ISTH) major bleeding
Secondary endpoints | 30 days and 12 months
  All bleeding complications scored by the Bleeding Academic Research Consortium (BARC) classification
Secondary endpoints | 24 hours to 24 months
  Change in the RV-to-LV diameter ratio as measured by echocardiography
Secondary endpoints | 24 hours to 24 months
  Change in the systolic pulmonary artery pressure (sPAP) as measured by echocardiography
Secondary endpoints | 24 hours to 24 months
  Change in the Tricuspid annular plane systolic excursion (TAPSE) as measured by echocardiography
Secondary endpoints | 24 hours to 24 months
  Change in the Tissue Doppler imaging-derived Tricuspid lateral annular Systolic Velocity (S´ TDI) as measured by echocardiography
Secondary endpoints | Discharge, 30 days, 12 months and 24 months
  Functional status as measured by World Health Organization (WHO) functional class
Secondary endpoints | 12 and 24 months
  Functional status as measured by the 6-Minute Walk Test (6MWT)
Secondary endpoints | 30 days to 24 months
  Quality of life using EuroQol-5D scale. The scale is numbered 0-100 with the value of 100 indicating the best health and the value of 0 indicating the worst health one can imagine
Secondary endpoints | 24 months
  Diagnosis of chronic thromboembolic pulmonary hypertension (CTEPH)

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Kocka, MD, PhD, Principal Investigator — Deputy Head of Department of Cardiology; Josef Kroupa, MD, PhD, Principal Investigator — Interventional Cardiologist
Locations (1):
- University Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
will need to follow local and EU GDPR valid at the completion time
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Becattini C, Agnelli G, Lankeit M, Masotti L, Pruszczyk P, Casazza F, Vanni S, Nitti C, Kamphuisen P, Vedovati MC, De Natale MG, Konstantinides S. Acute pulmonary embolism: mortality prediction by the 2014 European Society of Cardiology risk stratification model. Eur Respir J. 2016 Sep;48(3):780-6. doi: 10.1183/13993003.00024-2016. Epub 2016 May 12. PMID 27174887
- [Background] Steering Committee. Single-bolus tenecteplase plus heparin compared with heparin alone for normotensive patients with acute pulmonary embolism who have evidence of right ventricular dysfunction and myocardial injury: rationale and design of the Pulmonary Embolism Thrombolysis (PEITHO) trial. Am Heart J. 2012 Jan;163(1):33-38.e1. doi: 10.1016/j.ahj.2011.10.003. PMID 22172434
- [Background] Meyer G, Vicaut E, Danays T, Agnelli G, Becattini C, Beyer-Westendorf J, Bluhmki E, Bouvaist H, Brenner B, Couturaud F, Dellas C, Empen K, Franca A, Galie N, Geibel A, Goldhaber SZ, Jimenez D, Kozak M, Kupatt C, Kucher N, Lang IM, Lankeit M, Meneveau N, Pacouret G, Palazzini M, Petris A, Pruszczyk P, Rugolotto M, Salvi A, Schellong S, Sebbane M, Sobkowicz B, Stefanovic BS, Thiele H, Torbicki A, Verschuren F, Konstantinides SV; PEITHO Investigators. Fibrinolysis for patients with intermediate-risk pulmonary embolism. N Engl J Med. 2014 Apr 10;370(15):1402-11. doi: 10.1056/NEJMoa1302097. PMID 24716681
- [Background] Kuo WT, Banerjee A, Kim PS, DeMarco FJ Jr, Levy JR, Facchini FR, Unver K, Bertini MJ, Sista AK, Hall MJ, Rosenberg JK, De Gregorio MA. Pulmonary Embolism Response to Fragmentation, Embolectomy, and Catheter Thrombolysis (PERFECT): Initial Results From a Prospective Multicenter Registry. Chest. 2015 Sep;148(3):667-673. doi: 10.1378/chest.15-0119. PMID 25856269
- [Background] Piazza G, Hohlfelder B, Jaff MR, Ouriel K, Engelhardt TC, Sterling KM, Jones NJ, Gurley JC, Bhatheja R, Kennedy RJ, Goswami N, Natarajan K, Rundback J, Sadiq IR, Liu SK, Bhalla N, Raja ML, Weinstock BS, Cynamon J, Elmasri FF, Garcia MJ, Kumar M, Ayerdi J, Soukas P, Kuo W, Liu PY, Goldhaber SZ; SEATTLE II Investigators. A Prospective, Single-Arm, Multicenter Trial of Ultrasound-Facilitated, Catheter-Directed, Low-Dose Fibrinolysis for Acute Massive and Submassive Pulmonary Embolism: The SEATTLE II Study. JACC Cardiovasc Interv. 2015 Aug 24;8(10):1382-1392. doi: 10.1016/j.jcin.2015.04.020. PMID 26315743
- [Background] Kucher N, Boekstegers P, Muller OJ, Kupatt C, Beyer-Westendorf J, Heitzer T, Tebbe U, Horstkotte J, Muller R, Blessing E, Greif M, Lange P, Hoffmann RT, Werth S, Barmeyer A, Hartel D, Grunwald H, Empen K, Baumgartner I. Randomized, controlled trial of ultrasound-assisted catheter-directed thrombolysis for acute intermediate-risk pulmonary embolism. Circulation. 2014 Jan 28;129(4):479-86. doi: 10.1161/CIRCULATIONAHA.113.005544. Epub 2013 Nov 13. PMID 24226805
- [Background] Tapson VF, Sterling K, Jones N, Elder M, Tripathy U, Brower J, Maholic RL, Ross CB, Natarajan K, Fong P, Greenspon L, Tamaddon H, Piracha AR, Engelhardt T, Katopodis J, Marques V, Sharp ASP, Piazza G, Goldhaber SZ. A Randomized Trial of the Optimum Duration of Acoustic Pulse Thrombolysis Procedure in Acute Intermediate-Risk Pulmonary Embolism: The OPTALYSE PE Trial. JACC Cardiovasc Interv. 2018 Jul 23;11(14):1401-1410. doi: 10.1016/j.jcin.2018.04.008. PMID 30025734
- [Background] Avgerinos ED, Jaber W, Lacomis J, Markel K, McDaniel M, Rivera-Lebron BN, Ross CB, Sechrist J, Toma C, Chaer R; SUNSET sPE Collaborators. Randomized Trial Comparing Standard Versus Ultrasound-Assisted Thrombolysis for Submassive Pulmonary Embolism: The SUNSET sPE Trial. JACC Cardiovasc Interv. 2021 Jun 28;14(12):1364-1373. doi: 10.1016/j.jcin.2021.04.049. PMID 34167677
- [Background] Klein AJ, Shishehbor MH. Ultrasound-assisted catheter directed therapy (CDT) for pulmonary embolism versus standard CDT: Sounds of a cry for data! Vasc Med. 2019 Jun;24(3):248-250. doi: 10.1177/1358863X19838346. Epub 2019 Mar 27. No abstract available. PMID 30915915
- [Background] Kroupa J, Buk M, Weichet J, Malikova H, Bartova L, Linkova H, Ionita O, Kozel M, Motovska Z, Kocka V. A pilot randomised trial of catheter-directed thrombolysis or standard anticoagulation for patients with intermediate-high risk acute pulmonary embolism. EuroIntervention. 2022 Oct 7;18(8):e639-e646. doi: 10.4244/EIJ-D-21-01080. PMID 35620984
- [Background] Klok FA, Piazza G, Sharp ASP, Ni Ainle F, Jaff MR, Chauhan N, Patel B, Barco S, Goldhaber SZ, Kucher N, Lang IM, Schmidtmann I, Sterling KM, Becker D, Martin N, Rosenfield K, Konstantinides SV. Ultrasound-facilitated, catheter-directed thrombolysis vs anticoagulation alone for acute intermediate-high-risk pulmonary embolism: Rationale and design of the HI-PEITHO study. Am Heart J. 2022 Sep;251:43-53. doi: 10.1016/j.ahj.2022.05.011. Epub 2022 May 16. PMID 35588898
- [Background] Galderisi M, Cosyns B, Edvardsen T, Cardim N, Delgado V, Di Salvo G, Donal E, Sade LE, Ernande L, Garbi M, Grapsa J, Hagendorff A, Kamp O, Magne J, Santoro C, Stefanidis A, Lancellotti P, Popescu B, Habib G; 2016-2018 EACVI Scientific Documents Committee; 2016-2018 EACVI Scientific Documents Committee. Standardization of adult transthoracic echocardiography reporting in agreement with recent chamber quantification, diastolic function, and heart valve disease recommendations: an expert consensus document of the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2017 Dec 1;18(12):1301-1310. doi: 10.1093/ehjci/jex244. PMID 29045589
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2015 Mar;16(3):233-70. doi: 10.1093/ehjci/jev014. PMID 25712077